CLINICAL TRIAL: NCT05775562
Title: Early Pulmonary Effects of Excursion Deep Diving with Closed-circuit Gas Recycling: SPIDD Study
Acronym: SPIDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 29BRC21.0273
Record Dates: First submitted 2022-12-14; First posted 2023-03-20 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Physiopathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diving arm (Other): The standard arm involves all participants in the study. Subjects will perform pre-dive and post-dive examinations to characterize the respiratory impact of deep water diving
  Interventions: Diagnostic Test: Pre and post dive examinations

INTERVENTIONS:
Diagnostic Test: Pre and post dive examinations — Performing pre-dive examinations:
  - EFR by plethysmography cabin
  Realization of the examinations the day of the dive:
  * Portable Spirometry
  * Pulmonary ultrasound
  * Cardiac ultrasound
  * Measurement of circulating bubbles
  * ECG
  * Venous blood sampling (biological collection)
  * Water balance (Δweight/water intake)
  * EFR by plethysmography cabin
  * Weight measurement
  Realization of the examinations the day after the dive:
  * Venous blood sample (biological collection)
  * Portable Spirometry
  * Pulmonary ultrasound
  * Cardiac ultrasound
  * Weight measurement

SUMMARY:
Scuba diving with closed circuit gas rebreathers is currently booming. Initially developed for professional and military diving, this type of diving has become very successful in recreational activities.

The possibilities offered by this equipment are immense and reduce the constraints of exploration time and depth. More and more divers are seeking to reach depths previously considered unusual or inaccessible in recreational diving, beyond 100 meters. By pushing back these limits, the diver is exposed to new risks which should lead to a reflection on the means of prevention and treatment in case of incident.

The physiological repercussions of these deep dives are not well known. During daily deep excursions in the 90-120 meter zone, there is a significant reduction in vital capacity on leaving the dive, which persists and worsens the following day.

It seems necessary to confirm the importance of this impairment, never documented before, and to explore its mechanisms. A better knowledge of this respiratory impact could allow to improve the prevention and the preliminary evaluation of the medical aptitude of these divers.

ELIGIBILITY:
Inclusion Criteria:

* Diver ≥ 18 years old
* Recreational rebreather diver with a recognised qualification (Mixed Gas CCR training or equivalent) and the necessary experience for this type of diving who has scheduled a dive in the 60 metre depth zone
* Diver using his/her own equipment, i.e. a closed circuit rebreather with back lungs meeting CE standards.
* Having a medical certificate of no contraindication to the practice of underwater activities < 1 year issued by an authorised doctor
* Having taken out personal insurance covering this type of activity
* Voluntary and having given his/her express, free and informed consent
* Affiliated to the Social Security

Exclusion Criteria:

* Diver refusal
* Known previous respiratory pathology
* Use of medication that may alter pulmonary and/or vascular function as well as inflammatory and haemostasis parameters
* Any temporary contraindication to the practice of scuba diving
* Patient under guardianship or trusteeship
* Immersion beyond 30 metres within 7 days or any scuba diving within the previous 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Variation in Vital Capacity Measurement before and after diving | Day 0 (before diving)
  Vital capacity measurement will be performed by plethysmography and spirometry (Measurement of mobilizable and non-mobilizable lung volumes (mL))
Variation in Vital Capacity Measurement before and after diving | Day 0 (after diving)
  Vital capacity measurement will be performed by plethysmography and spirometry (Measurement of mobilizable and non-mobilizable lung volumes (mL))
Variation in Vital Capacity Measurement before and after diving | Day +1
  Vital capacity measurement will be performed by plethysmography and spirometry (Measurement of mobilizable and non-mobilizable lung volumes (mL))

SECONDARY OUTCOMES:
Variations in Spirometry data before and after diving | Day -XX before diving
  Measurement of SPO2 (%), CVF (L), VEMS (L), VEMS/CVF (%), DEP (L/S) and DEMM (L/S) before and after diving by spirometry
Variations in Spirometry data before and after diving | Day 0 (before diving)
  Measurement of SPO2 (%), CVF (L), VEMS (L), VEMS/CVF (%), DEP (L/S) and DEMM (L/S) before and after diving by spirometry
Variations in Spirometry data before and after diving | Day 0 (after diving)
  Measurement of SPO2 (%), CVF (L), VEMS (L), VEMS/CVF (%), DEP (L/S) and DEMM (L/S) before and after diving by spirometry
Variations in Spirometry data before and after diving | Day +1
  Measurement of SPO2 (%), CVF (L), VEMS (L), VEMS/CVF (%), DEP (L/S) and DEMM (L/S) before and after diving by spirometry
Variations in plethysmography data before and after diving | Day -XX before Day 0
  Measurement of CV max (L), CVF (L), VRE (L), VRI (L), VT (L), VEMS (L), VR (L) and CPT (L) before and after diving by plethysmography
Variations in plethysmography data before and after diving | Day -XX before Day 0
  Measurement of DEP (L.S), DEM 75 (L/S), DEM 50 (L/s), DEM 25 (L/S) before and after diving by plethysmography
Variations in plethysmography data before and after diving | Day 0 (before diving)
  Measurement of CV max (L), CVF (L), VRE (L), VRI (L), VT (L), VEMS (L), VR (L) and CPT (L) before and after diving by plethysmography
Variations in plethysmography data before and after diving | Day 0 (before diving)
  Measurement of DEP (L.S), DEM 75 (L/S), DEM 50 (L/s), DEM 25 (L/S) before and after diving by plethysmography
Variations in plethysmography data before and after diving | Day 0 (after diving)
  Measurement of CV max (L), CVF (L), VRE (L), VRI (L), VT (L), VEMS (L), VR (L) and CPT (L) before and after diving by plethysmography
Variations in plethysmography data before and after diving | Day 0 (after diving)
  Measurement of DEP (L.S), DEM 75 (L/S), DEM 50 (L/s), DEM 25 (L/S) before and after diving by plethysmography
Variations in plethysmography data before and after diving | Day +1
  Measurement of CV max (L), CVF (L), VRE (L), VRI (L), VT (L), VEMS (L), VR (L) and CPT (L) before and after diving by plethysmography
Variations in plethysmography data before and after diving | Day +1
  Measurement of DEP (L.S), DEM 75 (L/S), DEM 50 (L/s), DEM 25 (L/S) before and after diving by plethysmography
Variations in DLCO before and after diving | Day 0 (before diving)
  Measurement DLCO (mmol/(min*kPa) before and after diving
Variations in DLCO before and after diving | Day 0 (after diving)
  Measurement DLCO (mmol/(min*kPa) before and after diving
Variations in DLCO before and after diving | Day +1
  Measurement DLCO (mmol/(min*kPa) before and after diving
Variations in lung ultrasound (B lines) before and after diving | Day 0 (before diving)
  A B-line count should be performed, which is defined as vertical artefacts, mobile with breathing, continuous, originating from the pleural line and erasing the other artefacts. These artefacts indicate interstitial damage, the importance of which correlates with their number and a very good correlation with the quantity of extrapulmonary water.
Variations in lung ultrasound (B lines) before and after diving | Day 0 (after diving)
  A B-line count should be performed, which is defined as vertical artefacts, mobile with breathing, continuous, originating from the pleural line and erasing the other artefacts. These artefacts indicate interstitial damage, the importance of which correlates with their number and a very good correlation with the quantity of extrapulmonary water.
Variations in lung ultrasound (B lines) before and after diving | Day +1
  A B-line count should be performed, which is defined as vertical artefacts, mobile with breathing, continuous, originating from the pleural line and erasing the other artefacts. These artefacts indicate interstitial damage, the importance of which correlates with their number and a very good correlation with the quantity of extrapulmonary water.
Variations in lung ultrasound (condensations) before and after diving | Day 0 (before diving)
  Ultrasound signs of condensation or pleural effusions should be observed before and after diving.
Variations in lung ultrasound (condensations) before and after diving | Day 0 (after diving)
  Ultrasound signs of condensation or pleural effusions should be observed before and after diving.
Variations in lung ultrasound (condensations) data before and after diving | Day +1
  Ultrasound signs of condensation or pleural effusions should be observed before and after diving.
Variations in cardiac ultrasound pulmonary pressure (PAPs) before and after diving | Day 0 (before diving)
  Pulmonary arterial pressures are assessed by studying pulmonary artery Doppler flow (Acceleration Time) and right ventricular ejection time (RVET) and calculating the Acceleration/RVET ratio.
Variations in cardiac ultrasound pulmonary pressure (PAPs) before and after diving | Day 0 (after diving)
  Pulmonary arterial pressures are assessed by studying pulmonary artery Doppler flow (Acceleration Time) and right ventricular ejection time (RVET) and calculating the Acceleration/RVET ratio.
Variations in cardiac ultrasound pulmonary pressure (PAPs) before and after diving | Day +1
  Pulmonary arterial pressures are assessed by studying pulmonary artery Doppler flow (Acceleration Time) and right ventricular ejection time (RVET) and calculating the Acceleration/RVET ratio.
Variations in right ventricle function data before and after diving | Day 0 (before diving)
  Right ventricular systolic function is assessed by measuring the tricuspid annulus plane systolic excursion (TAPSE) in TM mode and calculating the LV shortening fraction.
Variations in right ventricle function data before and after diving | Day 0 (after diving)
  Right ventricular systolic function is assessed by measuring the tricuspid annulus plane systolic excursion (TAPSE) in TM mode and calculating the LV shortening fraction.
Variations in right ventricle function data before and after diving | Day +1
  Right ventricular systolic function is assessed by measuring the tricuspid annulus plane systolic excursion (TAPSE) in TM mode and calculating the LV shortening fraction.
Variations in decompression (circulating bubbles) data before and after diving | Day 0 (before diving)
  Detection of circulating bubbles by trans-thoracic ultrasound
Variations in decompression (circulating bubbles) data before and after diving | Day 0 (after diving)
  Detection of circulating bubbles by trans-thoracic ultrasound
Variations in biological markers of coagulation activation before and after diving | Day 0 (before diving)
  Measurement from the serum library (venous blood samples) of coagulation factors (TFPI, procoagulant microparticles, Fibrin monomer, PF4, C3a, C5a and platelet count) before and after diving. The analyses remain to be specified according to the results of other ongoing investigations
Variations in biological markers of coagulation activation before and after diving | Day 0 (after diving)
  Measurement from the serum library (venous blood samples) of coagulation factors (TFPI, procoagulant microparticles, Fibrin monomer, PF4, C3a, C5a and platelet count) before and after diving. The analyses remain to be specified according to the results of other ongoing investigations
Variations in biological markers of coagulation activation before and after diving | Day +1
  Measurement from the serum library (venous blood samples) of coagulation factors (TFPI, procoagulant microparticles, Fibrin monomer, PF4, C3a, C5a and platelet count) before and after diving. The analyses remain to be specified according to the results of other ongoing investigations
Variations in biomarkers of lipid peroxidation before and after diving | Day 0 (before diving)
  Measurement from the serum library (venous blood samples) of lipoperoxidation (F2-Isoprostane) before and after the dive. The analyses remain to be specified according to the results of other ongoing investigations.
Variations in biomarkers of lipid peroxidation before and after diving | Day 0 (after diving)
  Measurement from the serum library (venous blood samples) lipoperoxidation (F2-Isoprostane) before and after the dive. The analyses remain to be specified according to the results of other ongoing investigations.
Variations in biomarkers of lipid peroxidation before and after diving | Day +1
  Measurement from the serum library (venous blood samples) lipoperoxidation (F2-Isoprostane) before and after the dive. The analyses remain to be specified according to the results of other ongoing investigations.
Variations in biomarkers of oxidative stress before and after diving | Day 0 (before diving)
  Measurement from the serum library (venous blood samples) of oxidative stress factors before and after the dive. The analyses remain to be specified according to the results of other ongoing investigations.
Variations in biomarkers of oxidative stress before and after diving | Day 0 (after diving)
  Measurement from the serum library (venous blood samples) of oxidative stress factors before and after the dive. The analyses remain to be specified according to the results of other ongoing investigations.
Variations in biomarkers of oxidative stress before and after diving | Day +1
  Measurement from the serum library (venous blood samples) of oxidative stress factors (as F2-Isoprostane, 8-isoprostane) before and after the dive. The analyses remain to be specified according to the results of other ongoing investigations.
Variations in biological markers of inflammation before and after diving | Day 0 (before diving)
  Measurement of inflammation factors (CRP and IL1-β) from the serum library (venous blood samples) before and after the dive. The analyses remain to be specified according to the results of other ongoing investigations.
Variations in biological markers of inflammation before and after diving | Day 0 (after diving)
  Measurement of inflammation factors (CRP and IL1-β) from the serum library (venous blood samples) before and after the dive. The analyses remain to be specified according to the results of other ongoing investigations.
Variations in biological markers of inflammation before and after diving | Day +1
  Measurement of inflammation factors (CRP and IL1-β) from the serum library (venous blood samples) before and after the dive. The analyses remain to be specified according to the results of other ongoing investigations.
Variations in water balance before and after diving | Day 0 (before diving)
  Pre- and post-dive water intakes are quantified but no intake restrictions are requested : Weight measured by electronic scale (in kg)
Variations in water balance before and after diving | Day 0 (after diving)
  Pre- and post-dive water intakes are quantified but no intake restrictions are requested : Weight measured by electronic scale (in kg)
Variations in water balance before and after diving | Day +1
  Pre- and post-dive water intakes are quantified but no intake restrictions are requested : Weight measured by electronic scale (in kg)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de BREST, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.